CLINICAL TRIAL: NCT02467335
Title: Single-dose Pharmacokinetics of BMS-626529, Administered as BMS-663068, in Subjects With Hepatic Impairment Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 206280; AI438-053 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2015-05-20; First posted 2015-06-10 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir

ARMS (4):
- Healthy Subjects (Active Comparator): Healthy subjects will receive a single, oral dose of BMS-663068 on Day 1.
  Interventions: Drug: BMS-663068
- Hepatic Impaired Subjects - Mild Rating (Active Comparator): Mildly impaired subjects will receive a single, oral dose of BMS-663068 on Day 1.
  Interventions: Drug: BMS-663068
- Hepatic Impaired Subjects - Moderate Rating (Active Comparator): Moderately impaired subjects will receive a single, oral dose of BMS-663068 on Day 1.
  Interventions: Drug: BMS-663068
- Hepatic Impaired Subjects - Severe Rating (Active Comparator): Severly impaired subjects will receive a single, oral dose of BMS-663068 on Day 1.
  Interventions: Drug: BMS-663068

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068

SUMMARY:
A single oral dose study in subjects with hepatic impairment and healthy control subjects. Subjects will stay at the clinical facility where interval blood samplings will be obtained and examined for drug effect.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 18 to 70 years, inclusive
* BMI: 18.5 to 38 kg/m2
* Body weight great or equal to 45.5 kg
* Subjects with hepatic impairment
* Subjects with hepatic impairment must be on a stable dose of medication and/or treatment regimen
* Healthy subjects to the extent possible matched to the first four subjects with hepatic impairment with regard to age, body weight, and sex, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Exclusion Criteria:

* Any major surgery within 4 weeks of study drug administration
* Donation of blood to a blood bank or in a clinical study (except a screening visit) within 4 weeks of study drug administration (within 2 weeks for plasma only)
* Subject has required additional medication for hepatic encephalopathy within 12 months (6 months for severe hepatic impairment) prior to dosing
* Presence of severe ascites or edema in subjects, as judged by the PI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2015-10-03 (Actual); Study Completion 2015-10-03 (Actual)

PRIMARY OUTCOMES:
The effects of hepatic impairment on the single-dose peak plasma concentration Cmax of BMS-626529 (metabolite). | 5 days
The effects of hepatic impairment on the single-dose area under the plasma concentration versus time curve AUC (INF) of BMS-626529 (metabolite). | 5 days
The effects of hepatic impairment on the single-dose area under the plasma concentration versus time curve AUC (0-T) of BMS-626529 (metabolite). | 5 days

SECONDARY OUTCOMES:
The safety and tolerability of a 600-mg single dose of BMS-663068 in subjects with hepatic impairment and in healthy subjects through analysis of adverse events. | 5 days
  Adverse events will be arranged by system organ class, preferred term and hepatic function group. In addition, electrocardiogram readings will be summarized by time point relative to hepatic function group, and investigator-identified abnormalities, if present, will be listed.
The relationship between the Child-Pugh classification (including its components) as well as liver function tests and BMS-626529 profile PK parameters. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Hamilton, New Jersey, United States